CLINICAL TRIAL: NCT07005817
Title: Ameliorating Social Isolation: Identifying Factors That Impede or Facilitate Health-related Social Behavior Change
Brief Title: Keep Social Study for Young Adults
Acronym: KSSYA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-1184; 1R01MD018492-01 (NIH)
Record Dates: First submitted 2025-05-14; First posted 2025-06-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-05

CONDITIONS: Social Isolation; Loneliness
Keywords: Keep Social; Online; Young Adult
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: Our main models use longitudinal structural equation modeling, multilevel structural equation modeling, and regression analysis. Further details are provided in the statistical analysis plan.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Participants are exposed to a brief psychoeducational video, guided instructions for creating if-then behavioral plans, a simulated social media platform with background content, and target messages within the platform that encourage in-person social interactions with strangers and acquaintances.
  Interventions: Behavioral: Experimental Health Communication
- Placebo Control Arm (Placebo Comparator): Participants are exposed to a simulated social media platform with background content.
  Interventions: Behavioral: Simulated Social Media Platform Only

INTERVENTIONS:
Behavioral: Experimental Health Communication — Participants view a brief psychoeducational video about the value of connecting in-person with others and receive guided instructions for creating if-then behavioral plans for increasing moments of high-quality social connection. Over the next four weeks, they view messages on a simulated social media platform to encourage in-person, connections with strangers and acquaintances on a platform called Invibe. The Invibe feed will also have approximately 15 background posts each day from "users'" about their lives, including food, fitness, pets, and travel, common on social media platforms.
  During the 4-week Invibe phase, after participants complete each Day Report, they will view the Invibe simulated social media feed. Participant exposure to each target message will be both passive, via that day's feed, and forced, via inclusion on the Day Report. Participants will see 12 social media messages during this 4-week phase, shown in random order within the first 3 daily posts.
  Other Names: Educational Video, Simulated Social Media Platform, and Target Messages
  Arms: Experimental Arm
Behavioral: Simulated Social Media Platform Only — To rule out placebo and nonspecific effects, the Keep Social RCT engenders positive expectations in all participants by promoting the use of Invibe as a beta social media platform to build and maintain social ties, a framing that mirrors information-as-usual for wellness through social media connections. Those in the Placebo Control condition receive no further health communication (view no psychoeducational video) and encounter all background content on Invibe (all target messages excluded) with control posts that feature unrelated content.
  Other Names: Placebo Control Communication
  Arms: Placebo Control Arm

SUMMARY:
The Keep Social randomized control trial (RCT) is a 6-week, online study which will test whether, relative to a placebo control condition, an intervention that encourages high-quality in-person social interactions with strangers and acquaintances reduces young adults' (ages 18 - 29) social isolation and loneliness.

Participants will complete our 6-week protocol, which includes 6 weeks of passive ecological behavior sampling (i.e., geotracking) and Day Reports, our 4-week Invibe social media messages, plus recurrent Biweekly Assessments (BW1-BW4) that include both self-reported and behavioral measures. The first Monday following enrollment, participants complete the BW1 baseline survey to assess demographic characteristics and initial levels of all outcome variables (primary and secondary, ~20 min). They also (optionally) activate passive geotracking on this day and leave it activated, continuously, for the duration of the study.

During the 2-week baseline and 4-week Invibe phases, time-varying psychological and behavioral mediators and moderators will be assessed three times per week via Day Reports. To increase ecological validity, each week, two weekdays (i.e., Monday, Tuesday, Wednesday, or Thursday), and one weekend day (i.e., Friday, Saturday or Sunday) will be randomly selected. Day reports will not be assigned on Mondays if there is a biweekly assessment scheduled.

DETAILED DESCRIPTION:
Social isolation and its subjective counterpart loneliness-well established as risk factors for poor physical and mental health-have been rising at alarming rates in the US, especially among young adults. Mechanistic understanding of how best to build social connectedness to ameliorate social isolation is sorely needed to redirect life trajectories toward health and well-being. In creating this foundational knowledge, variations across individuals and geographic location merit focus because these variations may be associated with unique challenges and opportunities for initiating social interactions. The broad, overarching objective of this work is to conduct basic experimental research on social connectedness to test whether, how, where, and for whom health communication messages can motivate in-person interactions to reduce young adults' social isolation and loneliness. Our multi-disciplinary team brings together expertise in social psychology, emotion science, communication science, and public health and will carry out a 6-week randomized controlled trial-the Keep Social RCT-using our innovative and ecologically valid simulated social media platform and a suite of rigorous repeated measures of social behavior, loneliness, and other health relevant outcomes.

This program of research is designed to meet three specific aims. SPECIFIC AIM 1 is to use optimized health messages about the value of social connectedness for young adults (ages 18-29) to conduct the Keep Social RCT to build a rich empirical platform. Initial empirical work has already used a human-centered process to design health communication messages that included peer imagery and stories and tested them in an online experiment with >700 young adults. Messages that received the highest ratings for encouraging in-person interactions in this online experiment were selected for the Keep Social RCT, which is placebo-controlled with behavioral and survey assessments repeated over six weeks. SPECIFIC AIM 2 is to analyze theory-driven mechanisms through which health communication messages in the Keep Social RCT may reduce young adults' social isolation and loneliness to identify intervention targets. This aim will be met with longitudinal statistical modeling to test whether and how the experimental health communication messages improve social connectedness. SPECIFIC AIM 3 is to extend data analyses of the Keep Social RCT to identify moderators of reduced social isolation and loneliness to identify where and for whom effects are largest. This aim will be met with advanced statistical modeling to illuminate the conditions under which our health communication messages most effectively ameliorate social isolation and loneliness in young adults. Taken together, this research will provide a framework to identify intervention targets to guide subsequent translational work undertaken to reduce loneliness that has been increasing across the US.

ELIGIBILITY:
Inclusion Criteria:

* Use social media
* Own a smartphone
* Reside in urban or suburban regions
* Meet one or more criteria for membership in a sociodemographic population with increased risk of adverse health outcomes in the U.S.: at least 500 participants who identity as Black or African American, at least 500 participants who identify as Hispanic, at least 500 participants with low subjective social status - i.e., who report a 5 or lower on the MacArthur Subjective Social Status (SSS) ladder). Groupings are not mutually exclusive.

Exclusion Criteria:

* Reside in rural region

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1900 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Quantity of locations visited as a potential indicator of social opportunity | Continuous over the duration of the 6-week study
  Participants will be asked to download a geolocation app to their smartphone that tracks their physical location throughout the study. Number of locations visited is a count variable (integers), with a lower bound of zero and an upper bound to be determine by participant behavior.
Roaming entropy as a potential indicator of social opportunity | Continuous over the duration of the 6-week study
  Based on GPS data (i.e., coordinates and timestamps), roaming entropy (RE) scores are computed with RE higher for days where one visits a greater number of locations and exhibits greater uniformity in the time distribution across visited locations. A minimum RE value would be achieved by spending all day in a single location, whereas maximum RE would, theoretically, be achieved by spending an equal proportion of the day in each unique location in an environment. Possible range is 0.00 to 1.00; range in past datasets is 0.00 to 0.52.
Loneliness, Self-Report (Biweekly) | Baseline/Week 0, Week 2, Week 4, and Week 6
  Four items from the National Institute of Health (NIH) Toolbox Adult Social Relationship Scales with mean responses ranging from 1 to 5. Lower scores indicate reduced loneliness.
Loneliness, Self-Report (Day) | Included in Day Reports, 3 times a week, over the 6-week RCT
  One item: "Today, I felt lonely." Mean scores range from 1 to 7 with a lower score representing less loneliness.
Behavioral Motivational Value for Strangers-Smiling-with-Direct-Gaze | Week 4
  The behavioral measure of motivational value (a.k.a., Implicit Motivational Value, or iMV) is estimated in a choice task as k values for stimulus types using a reinforcement learning (RL) paradigm and computational approaches. The task stimuli include fractals that precede the presentation of headshot photos of unfamiliar others in the same age range as study participants. Those photos show persons with one of 3 facial expressions: smiling-with-direct-gaze, smiling-with-gaze-averted, and neutral-with-gaze-averted. Participants are instructed to select their preferred fractal.
  Following work by Waugh et al. Computational a priori starting range: -1.5 to 1.5, with higher means representing more motivation to experience the image type (e.g., strangers-smiling-with-direct-gaze) relative to the middle category (i.e., strangers-smiling-with-gaze-averted).
Social Connection, Open Text | Week 6
  Participants will respond to an open-ended writing prompt asking them to reflect on how socially connected (or not) they felt during the study.
  To index both loneliness and depression, both top-down (theory-driven) dictionary-based approaches, specifically the Linguistic Inquiry Word Count (LIWC) and also bottom-up (data-driven) open-vocabulary linguistic features (words, phrases, and topics) will be used. LIWC scores represent the relative frequency of designated words within each LIWC category, ranging from 0.0 to 1.0. Higher scores represent greater frequency of the designated word category.
  Latent Dirichlet Allocation modeling (LDA) will be used to generate "topics" that represent data-driven linguistic features. The investigators will compute the topic distribution of each participant, ranging from 0.0 to 1.0. Higher scores represent greater frequency of the designated topic.

SECONDARY OUTCOMES:
Anxiety, Self-Report | Baseline/Week 0, Week 2, Week 4, and Week 6
  4-item Patient Reported Outcomes Measurement Information System (PROMIS)-29 measure that assesses participants' frequency of experiencing symptoms of anxiety. As described in the statistical analysis plan, the investigators plan to use the anxiety measure as an indicator in a "negative mental health" latent variable. Mean scores range from 1 to 7 with a lower score representing less anxiety.
Depression, Self-Report | Baseline/Week 0, Week 2, Week 4, and Week 6
  4-item PROMIS-29 measure that assesses participants' frequency of experiencing symptoms of depression. As described in the statistical analysis plan, the investigators plan to use the depression measure as an indicator in a "negative mental health" latent variable. Mean scores range from 1 to 7 with a lower score representing fewer symptoms of depression.
Stress, Self-Report | Baseline/Week 0, Week 2, Week 4, and Week 6
  4-item PROMIS-29 measure that assesses participants' frequency of perceiving stress. As described in the statistical analysis plan, the investigators plan to use the measure of perceived stress as an indicator in a "negative mental health" latent variable. Mean scores range from 1 to 7 with a lower score representing decreased stress levels.
Flourishing Mental Health, Self-Report | Baseline/Week 0, Week 2, Week 4, and Week 6
  14 items from the Mental Health Continuum, Short Form (MHC-SF) assessing flourishing mental health (emotional, psychological, and social well-being). As described in the statistical analysis plan, the investigators plan to use the MHC-SF measure as an indicator in a "positive mental health" latent variable. Scale scores range from 0 to 4 with higher scores used as a proxy for "positive mental health".
Life Satisfaction, Self-Report | Baseline/Week 0, Week 2, Week 4, and Week 6
  5-item NIH PROMIS survey that assesses participants' frequency of experiencing satisfaction with their life from PROMIS v1.0 -General Life Satisfaction Short Form 5a. As described in the statistical analysis plan, the investigators plan to use the life satisfaction measure as an indicator in a "positive mental health" latent variable. Mean scores range from 1 to 7, with higher scores representing life satisfaction.
Belongingness, Self-Report | Baseline/Week 0, Week 2, Week 4, and Week 6
  12-item General Belongingness Scale which assesses participants' sense of belonging across multiple levels of social ties and an overall sense of belonging beyond all interpersonal relationships. Mean scores range from 1 to 7 with higher scores indicating a greater sense of belonging.
Alcohol Consumption | Week 2 and Week 6
  Four items from the CDC's Behavioral Risk Factor Surveillance System (BRFSS) assess the frequency and quantity, respectively, of participants' consumption of alcoholic drinks during the past 30 days. The average daily alcohol consumption is calculated by multiplying the number of drinking days per month, as reported by each drinker, by the average number of drinks consumed per drinking day by each drinker; and then the product of the average total number of drinks consumed by all drinkers is divided by 30 days.
Illness Symptoms, Self-Report | Included in Day Reports, 3 times a week, over the 6-week RCT
  Participants asked to report the extent to which they experienced illness symptoms on the day they took their survey using the following item: "Today, I felt physically unwell or under the weather." Mean scores range from 1 to 7, with higher scores representing a greater degree of illness.
Physical Pain, Self-Report | Included in Day Reports, 3 times a week, over the 6-week RCT
  One item asks participants the degree to which they felt impeded by bodily sensations of physical pain that day: "Today, I was bothered by physical pain." Mean scores range from 1 to 7, with higher scores indicating more pain.

OTHER OUTCOMES:
Motivation for Recommended Health Behavior | Week 2 (experimental group only)
  3 items adapted from the Person-Activity Fit Scale, which assesses the extent to which the recommended health behaviors fit with the participants' natural routine, bring enjoyment, and are valued, Experimental Group only.
  Measure: People do things for many different reasons. Thinking about this challenge to connect more often in-person with people you don't know (or hardly know), please rate why you might adopt this recommendation.
  * Because doing this activity will feel "natural" to me and I'll be able to stick with it.
  * Because I will enjoy doing it; I'll find it interesting and challenging.
  * Because I value and identify with doing it; I'll do it freely even when it's not enjoyable.
  Mean scores range from 1 to 7 and higher scores indicate participants willingness to adopt new behaviors.
Perceived Message Effectiveness, Self-Report | Included in Day Reports, 3 times a week, over the 6-week RCT
  One item to assess the extent to which the post motivates the intended behavior: "This post makes me want to connect in person with people I barely know more often." The mean score ranges from 1 to 7 and higher scores indicate higher motivation for the intended behavior.
Message Relevance, Self-Report | Included in Day Reports, 3 times a week, over the 6-week RCT
  One item to assess how relevant a given social media message is to the participant: "I can relate to the situation described in the post." The mean score ranges from 1 to 7 and higher scores indicate that the social media messages have more relevance to the participant.
Perceived Social Presence, Self-Report | Included in Day Reports, 3 times a week, over the 6-week RCT
  One item to assess how the extent to which a post creates feelings of being with others: "When viewing this post, I feel as if someone is talking to me." The mean score ranges from 1 to 7 with high scores indicating more social presence.
Behavioral Adherence, Self-Report | Included in Day Reports, 3 times a week, over the 6-week RCT
  Participants are first asked to report how often they were open to vs. initiated social contact with less familiar people: "Think back across the last few days and identify the most recent day that you were out and about. Answer the next questions about 'Today' with reference to that particular day." Item 1: "Today, when out and about, how often were you open to connecting with people you didn't know (or hardly knew)?" Item 2: "Today, when out and about, how often did you initiate connecting with people you didn't know (or hardly knew)?" Mean scores range from 1 to 5 with high scores indicating higher adherence.
Quantity of Social Interactions, Self-Report | Included in Day Reports, 3 times a week, over the 6-week RCT
  Participants are asked to report (in three separate questions) on the number of in-person social interactions that they had with three types of social ties in the previous 24 hours: strangers, less familiar people (e.g., neighbors, acquaintances, coworkers), and close others (e.g., friends, family members).
Emotional Quality of Social Interactions, Self-Report | Included in Day Reports, 3 times a week, over the 6-week RCT
  2 items from the Perceived Positivity Resonance Scale which assesses the degree to which participants' in-person social interactions that were characterized by a mutual sense of warmth, concern, and "in sync" with others. Positivity resonance with strangers, less familiar people, and close others are assessed separately. Participants are asked to recall a specific interaction within the last 24 hours with each type of tie (or within past few days if they did not have a social interaction with the relevant tie within the past 24 hours) and then report on the following two items: "During this interaction, to what extent did you experience a mutual sense of warmth and concern toward one another?" and "During this interaction, to what extent did you feel "in sync" with this person?" Mean scores range from 0 to 10, with higher values signaling more positivity resonance.
Positive Emotions, Explicit Self-Report | Included in Day Reports, 3 times per week, over the 6-week RCT
  Positive emotions are assessed using the following item: "Today I felt pleasant emotions (amusement, awe, gratitude, hope, inspiration, interest, joy, love, pride, or serenity.)" Mean scores range from 0 to 4, with higher scores indicating higher levels of positive emotion.
Perceived Incivility, Self-Report | Included in Day Reports, 3 times a week, over the 6-week RCT
  One item that asks participants to indicate the extent to which the following statement describes their day: "Today, someone put me down, was condescending to me, or otherwise disrespected me." Mean scores range from 1 to 7 with lower scores representing a lesser degree of incivility.
Prioritizing Positivity, Self-Report | Baseline/Week 0 and Week 6
  Five-item Prioritizing Positivity Resonance Scale which assesses the extent to which individuals seek positivity. Mean scores range from 1 to 9, with higher scores representing a greater degree of positivity.
Prioritizing Positivity Resonance, Self-Report | Baseline/Week 0 and Week 6
  One item assessing prioritizing in-person social connection "I structure my day to maximize quality in-person moments with people in general." Mean scores range from 1 to 9, with higher scores representing a greater degree of prioritizing in-person connections.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L. Frederickson, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed a data use/sharing agreement with UNC

REFERENCES:
- [Background] Catalino LI, Boulton AJ. The Psychometric Properties of the Prioritizing Positivity Scale. J Pers Assess. 2021 Sep-Oct;103(5):705-715. doi: 10.1080/00223891.2020.1828433. Epub 2020 Nov 9. PMID 33166185
- [Background] Hays RD, Spritzer KL, Schalet BD, Cella D. PROMIS(R)-29 v2.0 profile physical and mental health summary scores. Qual Life Res. 2018 Jul;27(7):1885-1891. doi: 10.1007/s11136-018-1842-3. Epub 2018 Mar 22. PMID 29569016
- [Background] Heller AS, Shi TC, Ezie CEC, Reneau TR, Baez LM, Gibbons CJ, Hartley CA. Association between real-world experiential diversity and positive affect relates to hippocampal-striatal functional connectivity. Nat Neurosci. 2020 Jul;23(7):800-804. doi: 10.1038/s41593-020-0636-4. Epub 2020 May 18. PMID 32424287
- [Background] Keyes CL, Wissing M, Potgieter JP, Temane M, Kruger A, van Rooy S. Evaluation of the mental health continuum-short form (MHC-SF) in setswana-speaking South Africans. Clin Psychol Psychother. 2008 May-Jun;15(3):181-92. doi: 10.1002/cpp.572. PMID 19115439
- [Background] Lim S, Cortina LM. Interpersonal mistreatment in the workplace: the interface and impact of general incivility and sexual harassment. J Appl Psychol. 2005 May;90(3):483-96. doi: 10.1037/0021-9010.90.3.483. PMID 15910144
- [Background] Major BC, Le Nguyen KD, Lundberg KB, Fredrickson BL. Well-Being Correlates of Perceived Positivity Resonance: Evidence From Trait and Episode-Level Assessments. Pers Soc Psychol Bull. 2018 Dec;44(12):1631-1647. doi: 10.1177/0146167218771324. Epub 2018 May 13. PMID 29756547
- [Background] Cyranowski JM, Zill N, Bode R, Butt Z, Kelly MA, Pilkonis PA, Salsman JM, Cella D. Assessing social support, companionship, and distress: National Institute of Health (NIH) Toolbox Adult Social Relationship Scales. Health Psychol. 2013 Mar;32(3):293-301. doi: 10.1037/a0028586. PMID 23437856
- [Background] Reneau TR, Villano WJ, Jaso BA, Heller AS. The affective benefits of real-world exploration during the COVID-19 pandemic. J Psychopathol Clin Sci. 2024 Feb;133(2):167-177. doi: 10.1037/abn0000888. Epub 2023 Dec 14. PMID 38095970
- [Background] Waugh CE, Porth AP, Fang X, Sands LP, Kishida KT. What do we actually want to experience? A computational metric for assessing reward values. Res Sq [Preprint]. 2025 Feb 17:rs.3.rs-5875678. doi: 10.21203/rs.3.rs-5875678/v1. PMID 40034432
- [Background] Lyubomirsky, S. The how of happiness: A scientific approach to getting the life you want. 2008. New York: Penguin Press
- [Background] Malone, GP, Pillow, DR, & Osman, A. The General Belongingness Scale (GBS): Assessing achieved belongingness. Personality and Individual Differences, 2012, 52(3), 311-316. https://doi.org/10.1016/j.paid.2011.10.027
- [Background] Salsman JM, Lai JS, Hendrie HC, Butt Z, Zill N, Pilkonis PA, Peterson C, Stoney CM, Brouwers P, Cella D. Assessing psychological well-being: self-report instruments for the NIH Toolbox. Qual Life Res. 2014 Feb;23(1):205-15. doi: 10.1007/s11136-013-0452-3. Epub 2013 Jun 16. PMID 23771709